CLINICAL TRIAL: NCT01723696
Title: Vitamin C to Decrease Effects of Smoking in Pregnancy on Infant Lung Function
Acronym: VCSIP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Office of Dietary Supplements (ODS) (NIH)
Responsible Party: Principal Investigator, Cynthia McEvoy, Associate Professor of Pediatrics, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HL105447; R01HL105447 (NIH)
Record Dates: First submitted 2012-11-06; First posted 2012-11-08 (Estimated); Results first posted 2019-04-17 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-03

CONDITIONS: Pulmonary Function; Newborn, Abnormal; Infant Wheeze; In-utero Nicotine; Second Hand Smoke
Keywords: In-utero smoke;; Pulmonary function testing;; Wheeze;; Vitamin C;; Forced expiratory flows
MeSH Terms: conditions — Antisocial Personality Disorder; Respiratory Sounds | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo tablet+prenatal vitamin (Placebo Comparator): A daily placebo tablet
  Interventions: Dietary Supplement: Placebo tablet+prenatal vitamin
- Vitamin C +prenatal vitamin (Active Comparator): 500 mg vitamin C /day
  Interventions: Dietary Supplement: Vitamin C +prenatal vitamin

INTERVENTIONS:
Dietary Supplement: Vitamin C +prenatal vitamin — Pregnant smoking women will be randomized to daily vitamin C (500 mg) versus daily placebo
  Other Names: Ascorbic acid
  Arms: Vitamin C +prenatal vitamin
Dietary Supplement: Placebo tablet+prenatal vitamin
  Arms: placebo tablet+prenatal vitamin

SUMMARY:
Vitamin C supplementation (500 mg per day) given to pregnant women who can not quit smoking will improve the pulmonary function tests in their offspring measured at 3 months of age.

DETAILED DESCRIPTION:
Smoking during pregnancy remains a major public health problem as at least 12% of pregnant women cannot quit smoking during pregnancy. This addiction is the largest preventable cause of childhood respiratory illness, including asthma, and children whose mothers smoked during pregnancy show lifetime decreases in pulmonary function. Smoking is a unique morbidity in that it is addictive, heavily advertised and recent genome studies show there are genotypes that significantly increase the likelihood of being unable to quit. Teen pregnancy, low income, low education, and living with another smoker are important factors increasing the odds of smoking during pregnancy. Pulmonary function tests done shortly after birth in babies born to mothers who smoked during pregnancy show decreased pulmonary function as measured by decreased respiratory flows and respiratory compliance and altered tidal breathing patterns. These changes can still be measured even after the infants have reached adulthood. Multiple epidemiologic studies show that these decreases in pulmonary function lead to increased respiratory disease and costs of hundreds of millions of dollars per year.

The primary aim of this double-blind, placebo controlled, randomized, multi-site study is to demonstrate improved pulmonary function testing at 3 months of age, in infants delivered to smoking mothers who are randomized to 500 mg/day of supplemental vitamin C versus placebo at less than or equal to 22 weeks of pregnancy. We will recruit 278 smoking pregnant women into the study. Patients will meet with research personnel at each prenatal visit and smoking cessation will be actively encouraged. Patients will be monitored with a set of serial biomarkers to assess smoking and medication compliance, including urine cotinine levels, smoking questionnaires, pill counts and fasting plasma ascorbic acid levels. Pulmonary function tests will be done at 3 months of age and will measure forced expiratory flows. The infants will also be followed through one year of age with monthly validated respiratory questionnaires and a follow-up pulmonary function test at 12 months of age. Success of this study is supported by strong pilot data showing statistically significant improvements at about 48 hours of age in pulmonary function tests in infants born to smoking mothers who received vitamin C versus placebo, and preliminary data showing a lower incidence of wheezing at 12 months of age in these infants. Key genetic polymorphisms shown to increase sensitivity to in-utero smoke exposure will also be measured. The success of this study is also supported by animal models showing the effectiveness of vitamin C to preserve pulmonary function and genetic and epidemiologic studies linking the effects of smoking during pregnancy to oxidant mechanisms. The secondary aims of the study include: 1) to demonstrate a decreased incidence of wheezing through 12 months of age in infants delivered to smoking mothers who are randomized to 500mg/day of supplemental vitamin C versus placebo during pregnancy; 2) to demonstrate improved pulmonary function tests at 12 months of age in these infants.

ELIGIBILITY:
Inclusion Criteria: At randomization:

* Singleton gestation
* ≥ 15 years old
* Gestational age between 13 and 22 weeks
* Receiving prenatal care
* Current smoker
* English speaking

Exclusion Criteria:

* Gestational age ≥ 23 and 0/7 weeks
* Multiple gestation
* Major fetal congenital anomalies
* Current use of illicit drugs
* Current alcohol abuse
* Use of vitamin C (≥ 500 mg/day)>3 days per week since last menstrual period
* Refusal to abstain from vitamin or supplements containing significant vitamin C other than those provided through or approved by study staff
* History of kidney stone in patient
* Insulin dependent diabetes
* Complex maternal medical conditions
* Participation in other conflicting research projects
* Unable to demonstrate stable method of communication
* Pregnancy by in-vitro fertilization
* Plan to terminate pregnancy
* Failure of medication compliance trial
* Failure to return in designated period during placebo run-in
* Body mass index > 50 at screening

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2012-12; Primary Completion 2016-04 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia T McEvoy, MD,MCR, Principal Investigator — Oregon Health and Science University
Locations (2):
- United States (2):
  - Indiana University, Indianapolis, Indiana
  - Oregon Health & Science University, Portland, Oregon

REFERENCES:
- [Derived] Shorey-Kendrick LE, McEvoy CT, Milner K, Harris J, Brownsberger J, Tepper RS, Park B, Gao L, Vu A, Morris CD, Thompson EE, Ober C, Spindel ER. Vitamin C supplementation to pregnant smokers alters asthma- and allergy-associated CpGs in child buccal DNA at 5 years of age. Clin Epigenetics. 2025 Oct 3;17(1):155. doi: 10.1186/s13148-025-01965-2. PMID 41044653
- [Derived] Shorey-Kendrick LE, McEvoy CT, Milner K, Harris J, Brownsberger J, Tepper RS, Park B, Gao L, Vu A, Morris CD, Spindel ER. Improvements in lung function following vitamin C supplementation to pregnant smokers are associated with buccal DNA methylation at 5 years of age. Clin Epigenetics. 2024 Feb 27;16(1):35. doi: 10.1186/s13148-024-01644-8. PMID 38413986
- [Derived] Shorey-Kendrick LE, McEvoy CT, O'Sullivan SM, Milner K, Vuylsteke B, Tepper RS, Haas DM, Park B, Gao L, Vu A, Morris CD, Spindel ER. Impact of vitamin C supplementation on placental DNA methylation changes related to maternal smoking: association with gene expression and respiratory outcomes. Clin Epigenetics. 2021 Sep 19;13(1):177. doi: 10.1186/s13148-021-01161-y. PMID 34538263
- [Derived] McEvoy CT, Shorey-Kendrick LE, Milner K, Schilling D, Tiller C, Vuylsteke B, Scherman A, Jackson K, Haas DM, Harris J, Schuff R, Park BS, Vu A, Kraemer DF, Mitchell J, Metz J, Gonzales D, Bunten C, Spindel ER, Tepper RS, Morris CD. Oral Vitamin C (500 mg/d) to Pregnant Smokers Improves Infant Airway Function at 3 Months (VCSIP). A Randomized Trial. Am J Respir Crit Care Med. 2019 May 1;199(9):1139-1147. doi: 10.1164/rccm.201805-1011OC. PMID 30522343

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study staff screened women at prenatal clinics between December, 2012 and June, 2015 in the catchment area of the three clinical sites to identify eligible women who continued to smoke cigarettes.
Pre-assignment Details: To exclude highly non-compliant subjects, consented patients entered a medication compliance trial of 14 ± 7 days. Placebo tablets were given to participants and they were excluded if they failed to return for a post compliance visit within 14 ± 7 days of the screening visit or if they took < 75% of the required tablets.
Groups:
- Placebo Tablet+Prenatal Vitamin: Participants in this arm were to take a daily placebo tablet+prenatal vitamin. Placebo tablets contained microcrystalline cellulose and 100 mg of citric acid to mimic the taste of Vitamin C.
Period: Overall Study
Arm/Group | Placebo Tablet+Prenatal Vitamin | Vitamin C +Prenatal Vitamin
Started | 126 | 126
Completed (Number of participants who completed the primary outcome.) | 109 | 113
Not Completed | 17 | 13

BASELINE CHARACTERISTICS:
Population: Baseline analysis population includes only 125 for the Vitamin C group because after randomization, it was discovered that one participant had violated the inclusion/exclusion criteria and the IRB required that their data be excluded from any analyses.
Groups:
- Placebo Tablet+Prenatal Vitamin: A daily placebo tablet
  Placebo tablet+prenatal vitamin
- Total: Total of all reporting groups
Arm/Group | Placebo Tablet+Prenatal Vitamin | Vitamin C +Prenatal Vitamin | Total
Number analyzed (Participants) | 126 | 125 | 251
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 6 | 16
  Between 18 and 65 years | 116 | 119 | 235
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.4 (5.9) | 26.6 (5.2) | 26.5 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126 | 125 | 251
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 2 | 9
  Not Hispanic or Latino | 119 | 122 | 241
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 15 | 20 | 35
  White | 100 | 97 | 197
  More than one race | 8 | 7 | 15
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 126 | 125 | 251
Marital Status [Count of Participants; unit: Participants]
  Married | 31 | 22 | 53
  Single | 49 | 39 | 88
  Divorced | 7 | 8 | 15
  Significant Other | 39 | 56 | 95
Highest Education Level Attained [Count of Participants; unit: Participants]
  Less than High School | 31 | 20 | 51
  High School or GED | 40 | 59 | 99
  Some College | 49 | 43 | 92
  Bachelor's Degree | 6 | 3 | 9
  Graduate School | 0 | 0 | 0
Health Insurance Type [Count of Participants; unit: Participants]
  Government Assistance | 106 | 112 | 218
  Private Insurance | 18 | 13 | 31
  None or Self Pay | 2 | 0 | 2
Gestational Age at Enrollment [Mean (Standard Deviation); unit: weeks] | 16.4 (2.9) | 16.7 (3.1) | 16.5 (3.0)
Gestational Age at Randomization [Mean (Standard Deviation); unit: weeks] | 18.2 (2.8) | 18.4 (3.0) | 18.3 (2.9)
BMI at Enrollment [Mean (Standard Deviation); unit: kg/m^2] | 30.0 (7.3) | 28.6 (6.5) | 29.3 (6.9)
Gravida [Mean (Standard Deviation); unit: pregnancies] | 3.5 (2.4) | 3.3 (2) | 3.4 (2.2)
Cigarette Smoking at Enrollment [Mean (Standard Deviation); unit: cigarettes per day] — This is the number of cigarettes mother reports smoking per day.
  cigarettes per day | 7.8 (4.9) | 8.0 (5.0) | 7.9 (4.9)
Cigarette Smoking 3 months prior to Pregnancy [Mean (Standard Deviation); unit: cigarettes per day] — Number of cigarettes mother reported smoking per day, 3 months prior to becoming pregnant
  cigarettes per day | 17.7 (10.8) | 15.9 (7.7) | 16.8 (9.4)
Maternal History of Asthma [Count of Participants; unit: Participants]
  Yes | 38 | 44 | 82
  No | 88 | 81 | 169
Maternal History of Substance Abuse [Count of Participants; unit: Participants]
  Yes | 16 | 20 | 36
  No | 110 | 105 | 215
Maternal History of Alcohol Abuse [Count of Participants; unit: Participants]
  Yes | 0 | 4 | 4
  No | 126 | 121 | 247

OUTCOME MEASURES:

1. Primary Outcome: Forced Expiratory Flow at 75% of Expired Volume (FEF75)
Description: The primary outcome was the comparison of infant FEFs at 3 months of age obtained using the raised volume rapid thoracic compression (RVRTC) technique in offspring of pregnant smokers randomized to vitamin C versus placebo. The specific primary outcome parameter was the measurement of FEF at 75% of the expired volume (FEF75)
Time Frame: 3 months of age
Population: Population included in analysis were infants who were able to complete technically acceptable PFT/FEF measurements at 3 months of age.
Measure: Mean (Standard Deviation); unit: ml/s
Arm/Group | Placebo Tablet+Prenatal Vitamin | Vitamin C +Prenatal Vitamin
Number analyzed (Participants) | 109 | 113
ml/s | 188.7 (66.4) | 200.7 (71.1)
Statistical Analysis 1: Comparison: Placebo Tablet+Prenatal Vitamin vs Vitamin C +Prenatal Vitamin; Our targeted sample size of 218 infants with successful FEFs at 3 months of age was determined to detect with 90% power, at a significance level of 0.05, increases of 15% in mean FEF75 in the vitamin C group compared to the placebo group; Test type: Superiority; p = 0.19, ANCOVA — P-value adjusted for design factors of site, gestational age at randomization and covariates of length, race, and sex of infant; Mean Difference (Final Values) = 12.1, 95% CI 2-sided [-6.1 to 30.3]

2. Secondary Outcome: Forced Expiratory Flow at 75% of Expired Volume (FEF75)
Description: The measurement of forced expiratory flows and specifically FEF75 will be done at 12 months of age in infants born to pregnant smoking women randomized to vitamin C versus placebo during pregnancy. FEF75 will be measured with the raised volume rapid thoracic compression technique.
Time Frame: 12 months of age
Population: These measurements were performed at the 12 month visit.
Measure: Mean (Standard Deviation); unit: mL/s
Arm/Group | Placebo Tablet+Prenatal Vitamin | Vitamin C +Prenatal Vitamin
Number analyzed (Participants) | 101 | 101
mL/s | 324 (84.1) | 351.6 (71.1)

3. Secondary Outcome: Incidence of Wheezing Through 12 Months of Age
Description: The incidence of wheezing through 12 months of age will be compared in the infants delivered to smoking pregnant women who were randomized to vitamin C (500 mg) versus placebo during pregnancy.
Time Frame: 12 months of age
Population: Population is infants who have reached 12 months of age, and whose parent/caregiver has completed at least 1 respiratory questionnaire past 122 days after birth.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Tablet+Prenatal Vitamin | Vitamin C +Prenatal Vitamin
Number analyzed (Participants) | 119 | 118
Participants | 63 | 51

ADVERSE EVENTS:
Time Frame: Adverse events were monitored and collect from time of enrollment until 12 months post delivery.
Description: Population at risk for infants are different than population at risk for mother/fetus because we had some dropout from time of randomization to delivery
Groups:
- Maternal/Fetal (Placebo): A daily placebo tablet
  Placebo tablet+prenatal vitamin
- Maternal/Fetal (Vitamin C): Vitamin C +prenatal vitamin: Pregnant smoking women will be randomized to daily vitamin C (500 mg) versus daily placebo
- Infant (Placebo): Infants of mothers in the Placebo group, who took a daily placebo + prenatal vitamin.
- Infant (Vitamin C): Infants of mothers in the Vitamin C group, who took daily vitamin C (500 mg) and a prenatal vitamin
Arm/Group | Maternal/Fetal (Placebo) | Maternal/Fetal (Vitamin C) | Infant (Placebo) | Infant (Vitamin C)
All-Cause Mortality (participants affected / at risk) | 1/126 | 1/125 | 1/123 | 1/120
Serious Adverse Events (participants affected / at risk) | 30/126 | 20/125 | 31/123 | 33/120
Other Adverse Events (participants affected / at risk) | 54/126 | 59/125 | 0/123 | 0/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maternal/Fetal (Placebo) (N=126) | Maternal/Fetal (Vitamin C) (N=125) | Infant (Placebo) (N=123) | Infant (Vitamin C) (N=120)
Syncope (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foetal heart rate deceleration (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Appendicitis perforated (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HELLP syndrome (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis ulcerative (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postpartum sepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anastomotic complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Convulsions (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Dysaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foetal growth restriction (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Placenta previa (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 10 (10) | 14 (14) | 0 (0) | 0 (0)
Premature labour (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 3 (4) | 2 (2) | 0 (0) | 0 (0)
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Threatened labour (Pregnancy, puerperium and perinatal conditions) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervical incompetence (Reproductive system and breast disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Endometritis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (6) | 0 (0) | 0 (0) | 1 (2)
Bronchitis viral (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endotracheal intubation (Surgical and medical procedures) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug withdrawal syndrome (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary valve stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Jaundice neonatal (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syndactyly (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Talipes (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyloric stenosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Congenital ureteric anomaly (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Congenital hydronephrosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skeletal dysplasia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Optic nerve hypoplasia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intussusception (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Duodenal atresia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fever neonatal (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Lethargy (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis neonatal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Convulsions (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia neonatal (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foetal exposure timing unspecified (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Necrotising enterocolititis neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 8 (8) | 9 (9)
Shoulder dystocia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug withdrawal syndrome neonatal (Psychiatric disorders) | 0 (0) | 0 (0) | 6 (6) | 3 (3)
Chordee (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Apparent life threatening event (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Cheyne-Stokes respiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metapneumovirus infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neonatal hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (5)
Cardio-respiratory arrest neonatal (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neonatal respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Respiratory syncytial virus bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Nephrectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Congenital aortic stenosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maternal/Fetal (Placebo) (N=126) | Maternal/Fetal (Vitamin C) (N=125) | Infant (Placebo) (N=123) | Infant (Vitamin C) (N=120)
Anaemia (Blood and lymphatic system disorders) | 9 (9) | 9 (9) | 0 (0) | 0 (0)
Gestational diabetes (Pregnancy, puerperium and perinatal conditions) | 16 (17) | 9 (11) | 0 (0) | 0 (0)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 19 (21) | 0 (0) | 0 (0)
Foetal hypokinesia (Pregnancy, puerperium and perinatal conditions) | 6 (6) | 7 (7) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 8 (8) | 16 (16) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Reproductive system and breast disorders) | 8 (8) | 12 (12) | 0 (0) | 0 (0)
Vaginitis bacterial (Reproductive system and breast disorders) | 9 (9) | 10 (10) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No